CLINICAL TRIAL: NCT06719492
Title: Development and Impact of a Nutrition Supplement and Nutrition Education on Patient Acceptance and Outcomes in Spine Surgery
Brief Title: Nutrition Education in Spine Surgery
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jennifer Bowden (Other)
Responsible Party: Sponsor-Investigator, Jennifer Bowden, Director of Research, Summit Brain,Spine,and Orthopedics
Organization: Summit Brain,Spine,and Orthopedics (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: SMI1351071
Record Dates: First submitted 2024-11-14; First posted 2024-12-05 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Nutrition Education; Enhanced Recovery After Surgery
MeSH Terms: interventions — Nutrition Assessment

STUDY DESIGN:
Intervention Model Description: One group receives additional nutrition education, the other (control) group receives typical clinic care. Both groups have an option to include a supplemental nutritional beverage if they choose.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nutrition education (Experimental): Participants randomized to this group will receive an additional 15 minutes of nutrition education focused on nutrition for surgical recovery. They will be offered an additional nutrition beverage if they choose it.
  Interventions: Behavioral: nutrition education
- Control group with typical clinic education and care (No Intervention): Participants randomized to this group will receive typical clinic education and care. They will be offered an additional nutrition beverage if they choose it.

INTERVENTIONS:
Behavioral: nutrition education — 15 minutes of surgery specific nutrition education provided by a Registered Dietitian.
  Arms: Nutrition education

SUMMARY:
The goal of this interventional study is to learn if having 15 minutes of surgery related nutrition education changes the food choices participants make during the time right before and after a spine surgery in participants who have a surgery with Dr. John Edwards. The main questions it aims to answer are:

* Does nutrition education at a participant's preoperative appointment help them choose healthier foods and drinks that help their recovery from surgery?
* Does choosing to drink some extra nutrients before and after surgery help participants feel better and make it easier to have other foods and liquids after surgery? Researchers will compare participants getting extra education with those in a control group who have normal instructions from the clinic to see if extra education makes a difference in people's food choices. Researchers will also look at how well participants do with the extra nutrition they get before and after surgery, and if choosing to include it changes with the extra education.

Participants will:

* Complete 2 surveys (PROMIS global and food frequency) at both their preoperative and postoperative appointments
* Complete one survey 2 days after their surgery asking about how well they did with liquids and solid foods in the 24 hours after surgery
* Choose whether or not they decide to have a drink with extra nutrients before and after surgery, and let the researchers know what they chose.

ELIGIBILITY:
Inclusion Criteria:

* Adult (18+ years of age)
* Patient of Dr. John Edwards undergoing spine surgery
* Patient is willing and able to complete all study requirements, including any education and follow up appointments

Exclusion Criteria:

* Under 18 years of age or pregnant
* Known allergies or intolerances to any supplement ingredients
* Patients deemed medically unstable by Dr. Edwards
* Patients with uncontrolled diabetes, as identified as Hemoglobin A1C>7.5
* Patients unwilling or unable to complete all study requirements including any education and follow up appointments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2024-11-05 (Actual); Primary Completion 2025-02-10 (Actual); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants in each group with changes in PROMIS global and food frequency questionnaire. | The study starts at the preoperative visit, typically 2 weeks prior to surgery, and ends at the first postoperative visit, which is typically 4 weeks after surgery for a total study duration of about 6-7 weeks.
  At both the preoperative and postoperative visits, participants will be given PROMIS Global and food frequency questionnaires.

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events of nausea and vomiting as assessed by CTCAE v4.0. | Total study duration is about 6-7 weeks from preoperative to initial postoperative visit, with this outcome measure being addressed 2 days following surgery.
  Nausea and vomiting and initial drinking and eating times will be evaluated comparing participants with extra nutrition education to those with standard care. Presence and severity of nausea and vomiting, and initial eating and drinking times by hours after surgery will be reported by participants 2 days after surgery in a texted survey.

OTHER OUTCOMES:
Participant satisfaction and learning as measured by change in food frequency questionnaire responses as well as time of initial food and liquid consumption after surgery. | The study starts at the preoperative visit, typically 2 weeks prior to surgery, and ends at the first postoperative visit, which is typically 4 weeks after surgery for a total study duration of about 6-7 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Bowden, PhD, RDN, Principal Investigator — Summit Brain,Spine,and Orthopedics
Locations (1):
- Summit Brain, Spine, and Orthopedics, Lehi, Utah, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hirsch KR, Wolfe RR, Ferrando AA. Pre- and Post-Surgical Nutrition for Preservation of Muscle Mass, Strength, and Functionality Following Orthopedic Surgery. Nutrients. 2021 May 15;13(5):1675. doi: 10.3390/nu13051675. PMID 34063333